CLINICAL TRIAL: NCT06737822
Title: Upfront Surgery Vs Induction Chemotherapy Followed By Surgery In Oral Cavity Squamous Cell Cancers With Advanced Nodal Disease (SurVIC Trial): A Phase 3 Multicentric Randomized Controlled Trial
Brief Title: Upfront Surgery Vs Induction Chemotherapy Followed By Surgery In Oral Cancers:
Acronym: SurVIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Jodhpur (Other Government)
Collaborators: All India Institute of Medical Sciences, Rishikesh (Other Government); All India Institute of Medical Sciences, Bhubaneswar (Other); All India Institute of Medical Sciences, Bathinda (Other Government); King George's Medical University (Other); Shri Mahant Indiresh Hospital, Dehradun (Unknown); Geetanjali Medical College, Udaipur (Unknown)
Responsible Party: Principal Investigator, Dharma Ram Poonia, Principal Investigator & Associate Professor Surgical Oncology, All India Institute of Medical Sciences, Jodhpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/5784
Record Dates: First submitted 2024-10-07; First posted 2024-12-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Oral Cancer; Head and Neck Neoplasms
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surg Arm (Active Comparator): Wide Local Excision (WLE) with Comprehensive neck dissection Adjuvant Treatment as per current standard Guidelines
  Interventions: Combination Product: Surgery and Adjuvant Treatment
- ICT Arm (Experimental): 2# of Chemotherapy before the Stadrard Surery: Either TPF or TPX Wide Local Excision (WLE) with Comprehensive neck dissection Adjuvant Treatment as per current standard Guidelines
  Interventions: Combination Product: TPF or TPX Regimen (2# ICT) --> Surgery and Adjuvant Treatment

INTERVENTIONS:
Combination Product: TPF or TPX Regimen (2# ICT) --> Surgery and Adjuvant Treatment — TPF:
  IINJ DOCETAXEL 75mg/M2 in 500 ML NORMAL SALINE(PVC free container/glass bottle) via codon filter OVER 60 MIN (DAY 1 ONLY) INJ. CISPLATIN 75 MG/M 2 IN 500 ML NS IV OVER 1 HOUR ON DAY1 ONLY INJ. 5FU 750 MG/M2 IV THROUGH INFUSION PUMP OVER 24 HOURS D 1-4
  Or
  TPX Regimen INJ DOCETAXEL 75mg/M2 in 500 ML NORMAL SALINE(PVC free container/glass bottle) via codon filter OVER 60 MIN (DAY 1 ONLY) INJ. CISPLATIN 75 MG/M 2 IN 500 ML NS IV OVER 1 HOUR ON D1 ONLY TAB. CAPECITABINE 850-1000MG/M2 TWICE A DAY 30 MINUTES AFTER MEALS FOR 14 DAYS IN A THREE WEEKLY CYCLE
  Surgery and Adjuvant Treatment Patients with PR/CR or SD will go for surgical resection. Patients having PD but still localized and resectable will be offered surgical resection, other would undergo radical CTRT or Palliative Treatment.
  Arms: ICT Arm
Combination Product: Surgery and Adjuvant Treatment — Wide Local Excision (WLE) with Comprehensive neck dissection and Adjuvant Treatment as per current standard Guidelines.
  Arms: Surg Arm

SUMMARY:
A majority of oral cancer patients in India present in the advanced stage hence tend to have poor oncological outcomes. Chemotherapy has been associated with improved oncological outcomes in various cancers but its role in oral cancer is not well defined in curative setting apart from radio sensitization. Attempted trials of neoadjuvant chemotherapy failed to show oncological advantage despite an excellent response rate, in part due to poor patient selection. Patients with a biologically aggressive disease are more likely to benefit, hence we intend to find out the oncological advantage of adding induction chemotherapy to oral squamous cell cancer with advanced nodal disease (N2-N3).

Earlier studies suffered from their heterogeneous patient population- all head and neck subsites together and included a spectrum ranging from early- stage operable cases to inoperable cancer. Due to such patient selection, the intended results were never met. The current study is intended to study the role of chemotherapy in curable patients who are most likely to benefit (biologically aggressive and advanced stage of presentation).

Objective

Primary:

To study the 2 year disease free survival by adding induction chemotherapy before surgery in patients of oral cancer with advanced nodal disease as compared to upfront surgery.

Secondary:

To assess treatment related outcomes between the treatment arms- Response rate; Treatment compliance; treatment related toxicity, postoperative complications and Quality of life.

To study the overall survival at 2 years. Oral cancer tissue biobanking for future translational research.

Study population Operable Oral cavity Squamous cell carcinoma with advanced nodal disease (N2-N3) Study Design Open label, Multi centric, randomized controlled trial with allocation ratio of 1:1

Sample Size The primary end point is disease-free survival. In order to have 80% power to detect a hazard ratio of 0.67, using a two-sided significance level, a total of 184 events are needed. Assuming an accrual rate of 15 patients a month, 300 patients need to be recruited. The analysis of DFS will take place 32 months after the start of the trial. The follow-up of patients will continue for 5 years. The analysis of OS will be conducted when 184 deaths are observed. taking 10% of withdrawal of consent, a total of 346 patients need to be included.

Inclusion Criteria Biopsy proven, operable oral Squamous cell carcinoma cT1-T4; cN2-N3, with adequate organ function, Age- 18-75 years, ECOG-PS:0-2 Treatment Arms

Standard Arm (SURG arm):

Surgery (Wide local Excision/composite resection with neck dissection) followed by adjuvant Radiotherapy ± Concurrent Chemotherapy

Experimental Arm (ICT):

2# TPF or TPX based induction chemotherapy followed by Surgery (Wide local Excision/composite resection with neck dissection) followed by adjuvant Radiotherapy ± Concurrent Chemotherapy

Study endpoints Primary- Disease free survival Secondary- Overall survival/ Quality of life/ Toxicity of treatment/ Treatment tolerance

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, treatment naïve, biopsy or cytology proven OSCC
* Clinical Stage cT1-4a, cN2-N3**, M0- as per UICC 2018
* No evidence of distant metastases on chest x-ray and/or CT Thorax
* ECOG PS 0-2
* No contraindication to Cisplatin or radiotherapy***
* Patients eligible for definitive curative intent treatment after discussion in multidisciplinary tumour board
* Adequate organ function at time of participation, defined as Haematological: Haemoglobin > 9gm/dl, ANC ≥ 1500/cmm3, Platelet ≥100000/cmm3 Liver Function test: Bilirubin ≤2 x upper limit normal (ULN), AST/ALT/ ALP ≤ 2.5 x ULN Renal Function test: Creatinine ≤ 1.5 ULN, Creatinine Clearance ≥60 ml/min.

Exclusion Criteria:

* Pregnant
* History of moderate to severe hearing loss.
* History of previous malignancy excluding non-melanoma skin cancers or cervical carcinoma in situ.
* Documented Weight loss of more than 15% in the last 6 months.
* Patients with known HIV, hepatitis B or C infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 2 Years
  Date of randomization to the date of clinical or pathological evidence of recurrence

SECONDARY OUTCOMES:
Overall Survival | 2 Years
  Date of randomization to the date of death due to any reason.
Treatment Completion Rate | 2 Years
  Number of Participants completing the treatment
Treatment Related Toxicity | 2 Years
  Chemotherapy Related and Radiotherapy Related: Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Quality of Life using PROs | 3 Months; 6 Months; 12 Months; 18 Months; 24 Months; 36 Months; 48 Months; 60 Months
  FACT HN Scale
Postoperative Surgical Morbidity | 30 Days and 90 Days
  Clavien Dindo Scale
Biobanking of Tumor, Non Tumor tissue and Blood | 2 Years
  DNA Sequencing using NGS to assess the genetic alterations
Financial Toxicity using Questionnaire | 3 Months; 6 Months; 12 Months; 18 Months; 24 Months; 36 Months; 48 Months; 60 Months
  FACT Scale
Early Radiotherapy Related Toxicity | 30 Days
  RTOG Criteria
Late Radiotherapy Relate Toxicity | 2 Years
  RTOG Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Dharma R Poonia, MS DNB, Principal Investigator — AIIMS Jodhpur
Locations (7):
- India (7):
  - All India Institute of Medical Sciences, Bhubaneshwar, Bhubaneshwar, Orisa
  - All India Institute of Medical Sciences, Jodhpur, Jodhpur, Rajasthan
  - All India Institute of Medical Sciences, Bathinda, Bathinda
  - Shri Mahant Indresh Hospital, Dehradun, Dehradun
  - King George's Medical University, Lucknow
  - All India Institute of Medical Sciences, Rishikesh, Rishikesh
  - Geetanjali Medical College, Udaipur, Udaipur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poonia DR, Sehrawat A, Vishnoi JR, Sharma N, Kumar P, Devnani B, Warriere A, Solanki A, Pareek P, Aggarwal D, Yadav T, Sharma PP, Gadwal A, Goyal A, Elhence P, Khera P, Jakhetiya A, Swaim P, Muduly D, Mahajan R, Garg P, Kumar V, Kar M, Misra S. Upfront surgery versus induction chemotherapy followed by surgery in oral cavity squamous cell cancers with advanced nodal disease (SurVIC Trial): a phase 3 multicentre randomised controlled trial. BMJ Open. 2025 Oct 6;15(10):e106644. doi: 10.1136/bmjopen-2025-106644. PMID 41057182